CLINICAL TRIAL: NCT06881316
Title: Caffeine vs. Carbohydrate Mouth Rinsing in Soccer: Effects on Passing Performance and Psychophysiological Responses in Youth Players
Brief Title: Caffeine vs. Carbohydrate Mouth Rinsing in Soccer
Acronym: CAFMR-CHOMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ersan Arslan, Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UGaziosmanpasa-1
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Performance; Soccer; Caffeine and Carbohydrate; Cognitive Function; Technical Skill
Keywords: Performance; caffeine mouth-rinsing; carbohydrate mouth-rinsing; cognitive-motor function; technical skill execution
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were strictly separated and think their intervention is the main intervention. The same was true for care providers. Outcome assessors were unaware of participant group status and were not allowed to ask correspondingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Caffeine Mouth Rinse Protocol (CAF-MR) (Experimental): Caffeine solutions (1.2% w/v caffeine solution) were prepared in an equivalent saccharin base to ensure indistinguishability within the Falcon Sterile Tube and agitated for 30 seconds on a vortex mixer. Participants were instructed to avoid intense activity 24 hours before testing, observe a 2-hour fast before sessions, and abstain from caffeinated products on test days. The following three sessions were test trials conducted between 15.00 h and 17.00 h at 32°C and 40% humidity.
  Interventions: Other: Caffeine
- CHO Mouth Rinse Protocol (CHO-MR) (Experimental): CHO solutions (6% w/v glucose solution) were prepared in an equivalent saccharin base to ensure indistinguishability within the Falcon Sterile Tube and agitated for 30 seconds on a vortex mixer. Participants were instructed to avoid intense activity 24 hours before testing, observe a 2- hour fast before sessions, and abstain from caffeinated products on test days. The following three sessions were test trials conducted between 15.00 h and 17.00 h at 32°C and 40% humidity.
  Interventions: Other: CHO
- Control Condition (Experimental): Only exercise was performed without any condition.
  Interventions: Other: Control

INTERVENTIONS:
Other: Caffeine — Participants' solutions were prepared in separate Falcon Sterile Tubes: LSPTCAFF (1.2% w/v caffeine solution, Nature's Supreme). An MRI was performed before the LSPT. The solution was sweetened with non-caloric artificial sweeteners consisting of sucralose. The caffeine solution was prepared in an equivalent saccharin base and shaken for 30 seconds in a vortex mixer to ensure distinguishability. Participants swished the solution in their mouth for 10 seconds before LSPT and then emptied it back into the container to be weighed again. To ensure that the solutions were not swallowed, the containers were measured before and after all MRs using a full precision balance (Etekcity, USA) accurate to 1 g/0.04 oz.
  Arms: Caffeine Mouth Rinse Protocol (CAF-MR)
Other: CHO — Participants' solutions were prepared in separate Falcon Sterile Tubes: LSPTCHO (6% w/ v glucose solution, Protein Ocean, Turkey) An MRI was performed prior to LSPT. The solution was sweetened with non-caloric artificial sweeteners consisting of sucralose. The CHO solution was prepared in an equivalent saccharin base and shaken for 30 seconds in a vortex mixer to ensure distinguishability. Participants swished the solution in their mouth for 10 seconds before LSPT and then emptied it back into the container to be weighed again. To ensure that the solutions were not swallowed, the containers were measured before and after all MRs using a full precision balance (Etekcity, USA) accurate to 1 g/0.04 oz.
  Arms: CHO Mouth Rinse Protocol (CHO-MR)
Other: Control — For the control condition, no supplements were taken and only exercise was performed.
  Arms: Control Condition

SUMMARY:
The present study evaluated the influence of carbohydrate mouth-rinsing (CHO-MR), caffeine mouth-rinsing (CAF-MR), and control-substance mouth rinses on Loughborough soccer passing test (LSPT) performance. The study participants were involved in a randomized, double-blind, repeated-measures design that employed four sessions (familiarization, CHOMR, CAFMR, and CONT) over ten days at a testing facility. Participants took part in six test sessions 72 hours apart. In the CHO group, 6% w/v glucose solution was used. In the CAFF group, 6% w/v glucose solution was used. CONT group, only exercise was performed without any condition.

DETAILED DESCRIPTION:
Participants were involved in a randomized, double-blind, repeated-measures design that employed four sessions (familiarization, LSPTCHO, LSPTCAFF, and LSPTCONT) over ten days at a testing facility. The initial session was an orientation, allowing participants to acclimate to the LSPT protocol and provide written informed consent. This session used water as a mouth rinse. Anthropometric data were also collected. Before the LSPT, participants completed 15-minute standardized warm-up sections, including jogging, sprinting, and integrating soccer-specific actions. The participants were asked to complete the LSPT at any time. During the tests, participants were blinded to the test scores. The following three sessions were test trials conducted between 15.00 h and 17.00 h at 32°C and 40% humidity. The participants performed the LSPT 72 h apart, LSPTCHO (6% w/v glucose solution), LSPTCAFF (1.2% w/v caffeine solution), and LSPTCONT conditions. Caffeine and CHO solutions were prepared in an equivalent saccharin base to ensure indistinguishability within the Falcon Sterile Tube and agitated for 30 seconds on a vortex mixer. Participants were instructed to avoid intense activity 24 hours before testing, observe a 2-hour fast before sessions, and abstain from caffeinated products on test days. All the test sessions were performed at 32°C and 40% humidity.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy
* Male soccer players
* Willing to maintain the intervention for all sessions

Exclusion Criteria:

* Being under 14 years old
* Having a chronic disease
* Contraindication for caffeine mouth-rinsing (CAF-MR)
* Contraindication for carbohydrate mouth-rinsing (CHO-MR)
* Contraindications for exercise

Ages: 14 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Psychophysiological Responses-Heart Rate | From baseline to the end of treatment at 2 weeks
  Participants used a Polar H10 heart rate (HR) transmitter synchronized with a Polar V800 watch to track the HR throughout the session. Participants' heart rate mean, heart rate peak and heart rate percentage were recorded.
Psychophysiological Responses-Rating of Perceived Exertion | From baseline to the end of treatment at 2 weeks
  Exercise intensity in all test sessions was quantified using the rating of perceived exertion (RPE), which employs a category ratio scale ranging from 6 to 20. This scale has recently been applied in sports psychology to assess effort related to emotions and performance during competitive events.
Psychophysiological Responses-Enjoyment-Brunel mood of states | From baseline to the end of treatment at 2 weeks
  all participants completed the exercise enjoyment scale (EES), which comprises eight items rated on a 1-7 Likert scale. This scale has been validated to measure enjoyment in Turkish adolescents and adults. To assess subjective mental fatigue levels, participants were instructed to indicate their degree of mental fatigue on a Visual Analog Scale (VAS).
Loughborough Soccer Passing Test (LSPT) | From baseline to the end of treatment at 2 weeks
  Participants were informed that the LSPT was a timed performance assessment and instructed to complete it as expeditiously as possible while minimizing penalties. The LSPT comprises 16 passes: eight short passes to red and white targets 3.5m from the passing zone and eight slightly longer passes to green and blue targets 4m away. Targets were constructed by affixing colored cards (0.3 x 0.6m) to the center of standard gymnasium benches, with a vertical aluminum strip (0.1 x 0.15m) fixed to the target's center for auditory feedback on successful passes. Four randomized passing sequences were generated. An examiner announces that the subsequent target color is released immediately after the previous pass. A stopwatch measured the test duration, commencing when the participant moved the ball into the passing zone and concluding when the final pass contacted the target area.

SECONDARY OUTCOMES:
Anthropometric Measurements 1 | Baseline
  Before breakfast, participants had their weight (kg) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.

OTHER OUTCOMES:
Anthropometric Measurements 2 | Baseline
  Before breakfast, participants had their height (cm) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.
Anthropometric Measurements 3 | Baseline
  Before breakfast, participants had their body mass index (kg/m2) measured using a body composition analyser (BC-418MA, Tanita Corp., Tokyo, Japan). This device utilises bioelectrical impedance technology using multiple frequencies (ranging from 1 kHz to 50 kHz) to comprehensively assess body composition parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Ersan Arslan, Doctorate, Study Chair — +905325452848
Locations (1):
- Tokat Gaziosmanpasa Universty, Tokat Province, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soylu Y, Ramazanoglu F, Arslan E, Clemente FM. Effects of mental fatigue on the psychophysiological responses, kinematic profiles, and technical performance in different small-sided soccer games. Biol Sport. 2022 Oct;39(4):965-972. doi: 10.5114/biolsport.2022.110746. Epub 2021 Dec 30. PMID 36247954
- [Background] Soylu Y, Chmura P, Arslan E, Kilit B. The Effects of Carbohydrate Mouth Rinse on Psychophysiological Responses and Kinematic Profiles in Intermittent and Continuous Small-Sided Games in Adolescent Soccer Players: A Randomized, Double-Blinded, Placebo-Controlled, and Crossover Trial. Nutrients. 2024 Nov 15;16(22):3910. doi: 10.3390/nu16223910. PMID 39599695